CLINICAL TRIAL: NCT01335464
Title: A 52 Weeks, Double Blind, Randomized, Placebo-controlled Trial Evaluating the Effect of Oral BIBF 1120, 150 mg Twice Daily, on Annual Forced Vital Capacity Decline, in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Safety and Efficacy of BIBF 1120 at High Dose in Idiopathic Pulmonary Fibrosis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1199.32; 2010-024251-87 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-04-13; First posted 2011-04-14 (Estimated); Results first posted 2015-02-13 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-06

CONDITIONS: Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis | interventions — nintedanib

ARMS (2):
- BIBF 1120 (Experimental): patient receives capsules containing BIBF 1120 twice a day
  Interventions: Drug: BIBF 1120
- placebo (Placebo Comparator): patient receives capsules identical to those containing active drug
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — placebo matching BIBF1120, BID
  Arms: placebo
Drug: BIBF 1120 — BIBF1120 BID (twice daily)
  Arms: BIBF 1120

SUMMARY:
Idiopathic Pulmonary Fibrosis (IPF) is a chronic disease of unknown cause that results in scarring of the lung and there is a high unmet medical need for effective treatment to halt lung function decline, delay or avoid exacerbation (flare-ups), and ultimately to reduce the death rate.

In a large Phase 2 trial (1199.30) (NCT00514683), investigating the effects of 52 weeks of treatment with BIBF 1120 in patients with IPF, a positive effect was seen on lung function of patients treated with high dose of BIBF 1120 compared to placebo.

Hence it is the purpose of this trial to investigate and confirm the efficacy and safety of BIBF 1120 at a high dose in treating patients with IPF, compared with placebo. The trial will be conducted as a prospective, randomised design with the aim to collect safety and efficacy data.

Respiratory function is globally accepted for assessment of treatment effects in IPF patients. The chosen endpoint (Forced Vital Capacity (FVC) decline) is easy to obtain and is part of the usual examinations done in IPF patients.

ELIGIBILITY:
Inclusion criteria:

1. Age >= 40 years;
2. IPF diagnosed, according to most recent American Thoracic Society (ATS), European Respiratory Society (ERS), Japanese Respiratory Society (JRS), Latin American Thoracic Association (ALAT) IPF guideline for diagnosis and management, within 5 years;
3. Combination of High Resolution Computerized Tomography (HRCT) pattern, and if available surgical lung biopsy pattern, as assessed by central reviewers, are consistent with diagnosis of IPF
4. Dlco (corrected for Hb): 30%-79% predicted of normal;
5. FVC>= 50% predicted of normal

Exclusion criteria:

1. Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) > 1.5 x Upper Limit of Normal (ULN)
2. Bilirubin > 1.5 x ULN;
3. Relevant airways obstruction (i.e. pre-bronchodilator FEV1/FVC < 0.7);
4. Patient likely to have lung transplantation during study (being on transplantation list is acceptable for participation);
5. Myocardial infarction within 6 months;
6. Unstable angina within 1 month;
7. Bleeding risk (genetic predisposition; fibrinolysis or full-dose therapeutic anticoagulation or high dose antiplatelet therapy; history of hemorrhagic CNS event within 12 months; haemoptysis or haematuria or active gastro-intestinal bleeding or ulcers or major injury or surgery within 3 months);
8. Thrombotic risk (inherited predisposition; history of thrombotic event (including stroke and transient ischemic attacks) within 12 months;
9. International normalised ratio (INR) > 2, prolongation of prothrombin time (PT) and partial thromboplastin time (PTT) by > 50% of institutional ULN);
10. N-ACetyl Cystein, prednisone > 15mg/day or equivalent received within 2 weeks of visit 1;
11. Pirfenidone, azathioprine, cyclophosphamide, cyclosporine A received within 8 weeks of visit 1;

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2011-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (98):
- United States (24):
  - 1199.32.10007 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1199.32.10029 Boehringer Ingelheim Investigational Site, Jasper, Alabama
  - 1199.32.10013 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 1199.32.10005 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1199.32.10022 Boehringer Ingelheim Investigational Site, Danbury, Connecticut
  - 1199.32.10025 Boehringer Ingelheim Investigational Site, Newark, Delaware
  - 1199.32.10023 Boehringer Ingelheim Investigational Site, Weston, Florida
  - 1199.32.10001 Boehringer Ingelheim Investigational Site, Council Bluffs, Iowa
  - 1199.32.10028 Boehringer Ingelheim Investigational Site, Wichita, Kansas
  - 1199.32.10016 Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - 1199.32.10024 Boehringer Ingelheim Investigational Site, New Brunswich, New Jersey
  - 1199.32.10019 Boehringer Ingelheim Investigational Site, New York, New York
  - 1199.32.10004 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1199.32.10020 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 1199.32.10002 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 1199.32.10033 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 1199.32.10008 Boehringer Ingelheim Investigational Site, Providence, Rhode Island
  - 1199.32.10015 Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - 1199.32.10034 Boehringer Ingelheim Investigational Site, Shelbyville, Tennessee
  - 1199.32.10009 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1199.32.10018 Boehringer Ingelheim Investigational Site, McKinney, Texas
  - 1199.32.10021 Boehringer Ingelheim Investigational Site, Falls Church, Virginia
  - 1199.32.10003 Boehringer Ingelheim Investigational Site, Lynchburg, Virginia
  - 1199.32.10038 Boehringer Ingelheim Investigational Site, Tacoma, Washington
- Australia (5):
  - 1199.32.61001 Boehringer Ingelheim Investigational Site, Camperdown, New South Wales
  - 1199.32.61002 Boehringer Ingelheim Investigational Site, Concord, New South Wales
  - 1199.32.61003 Boehringer Ingelheim Investigational Site, Daw Park, South Australia
  - 1199.32.61005 Boehringer Ingelheim Investigational Site, Frankston, Victoria
  - 1199.32.61004 Boehringer Ingelheim Investigational Site, Prahran, Victoria
- Belgium (4):
  - 1199.32.32004 Boehringer Ingelheim Investigational Site, Brussels
  - 1199.32.32005 Boehringer Ingelheim Investigational Site, Jette
  - 1199.32.32001 Boehringer Ingelheim Investigational Site, Leuven
  - 1199.32.32002 Boehringer Ingelheim Investigational Site, Yvoir
- China (6):
  - 1199.32.86001 Boehringer Ingelheim Investigational Site, Beijing
  - 1199.32.86002 Boehringer Ingelheim Investigational Site, Beijing
  - 1199.32.86005 Boehringer Ingelheim Investigational Site, Changsha
  - 1199.32.86004 Boehringer Ingelheim Investigational Site, Chengdu
  - 1199.32.86003 Boehringer Ingelheim Investigational Site, Nanchang
  - 1199.32.86006 Boehringer Ingelheim Investigational Site, Xi'an
- Czechia (3):
  - 1199.32.42002 Boehringer Ingelheim Investigational Site, Prague
  - 1199.32.42003 Boehringer Ingelheim Investigational Site, Prague
  - 1199.32.42001 Boehringer Ingelheim Investigational Site, Ústí nad Labem
- France (7):
  - 1199.32.33002 Boehringer Ingelheim Investigational Site, Bobigny
  - 1199.32.33003 Boehringer Ingelheim Investigational Site, Nice
  - 1199.32.33001 Boehringer Ingelheim Investigational Site, Paris
  - 1199.32.33005 Boehringer Ingelheim Investigational Site, Paris
  - 1199.32.33006 Boehringer Ingelheim Investigational Site, Paris
  - 1199.32.33007 Boehringer Ingelheim Investigational Site, Reims
  - 1199.32.33004 Boehringer Ingelheim Investigational Site, Rennes
- Germany (8):
  - 1199.32.49008 Boehringer Ingelheim Investigational Site, Bamberg
  - 1199.32.49005 Boehringer Ingelheim Investigational Site, Donaustauf
  - 1199.32.49001 Boehringer Ingelheim Investigational Site, Essen
  - 1199.32.49002 Boehringer Ingelheim Investigational Site, Freiburg/Breisgau
  - 1199.32.49006 Boehringer Ingelheim Investigational Site, Giessen
  - 1199.32.49003 Boehringer Ingelheim Investigational Site, Großhansdorf
  - 1199.32.49007 Boehringer Ingelheim Investigational Site, Heidelberg
  - 1199.32.49004 Boehringer Ingelheim Investigational Site, Mainz
- India (5):
  - 1199.32.91003 Boehringer Ingelheim Investigational Site, Ahmedabad
  - 1199.32.91002 Boehringer Ingelheim Investigational Site, Coimbatore
  - 1199.32.91006 Boehringer Ingelheim Investigational Site, Jaipur
  - 1199.32.91005 Boehringer Ingelheim Investigational Site, Kolkata
  - 1199.32.91001 Boehringer Ingelheim Investigational Site, Mumbai
- 1199.32.35301 Boehringer Ingelheim Investigational Site, Dublin, Ireland
- Israel (3):
  - 1199.32.97004 Boehringer Ingelheim Investigational Site, Haifa
  - 1199.32.97001 Boehringer Ingelheim Investigational Site, Petah Tikva
  - 1199.32.97002 Boehringer Ingelheim Investigational Site, Rehovot
- Italy (12):
  - 1199.32.39012 Boehringer Ingelheim Investigational Site, Catania
  - 1199.32.39004 Boehringer Ingelheim Investigational Site, Chieti Scalo
  - 1199.32.39008 Boehringer Ingelheim Investigational Site, Forlì
  - 1199.32.39005 Boehringer Ingelheim Investigational Site, Milan
  - 1199.32.39001 Boehringer Ingelheim Investigational Site, Modena
  - 1199.32.39007 Boehringer Ingelheim Investigational Site, Monza
  - 1199.32.39011 Boehringer Ingelheim Investigational Site, Napoli
  - 1199.32.39002 Boehringer Ingelheim Investigational Site, Padua
  - 1199.32.39006A Boehringer Ingelheim Investigational Site, Pisa
  - 1199.32.39006B Boehringer Ingelheim Investigational Site, Pisa
  - 1199.32.39010 Boehringer Ingelheim Investigational Site, Roma
  - 1199.32.39009 Boehringer Ingelheim Investigational Site, Siena
- Japan (12):
  - 1199.32.81005 Boehringer Ingelheim Investigational Site, Bunkyo-ku,Tokyo
  - 1199.32.81006 Boehringer Ingelheim Investigational Site, Bunkyo-ku,Tokyo
  - 1199.32.81007 Boehringer Ingelheim Investigational Site, Kiyose, Tokyo
  - 1199.32.81004 Boehringer Ingelheim Investigational Site, Kumagaya, Saitama
  - 1199.32.81009 Boehringer Ingelheim Investigational Site, Minato-ku, Tokyo
  - 1199.32.81003 Boehringer Ingelheim Investigational Site, Naka-gun, Ibaraki
  - 1199.32.81011 Boehringer Ingelheim Investigational Site, Ota-ku, Tokyo
  - 1199.32.81001 Boehringer Ingelheim Investigational Site, Sendai, Miyagi
  - 1199.32.81010 Boehringer Ingelheim Investigational Site, Shibuya-ku, Tokyo
  - 1199.32.81002 Boehringer Ingelheim Investigational Site, Shimotsuke,Tochigi
  - 1199.32.81008 Boehringer Ingelheim Investigational Site, Shinjuku-ku, Tokyo
  - 1199.32.81012 Boehringer Ingelheim Investigational Site, Yokohama, Kanagawa
- United Kingdom (8):
  - 1199.32.44006 Boehringer Ingelheim Investigational Site, Aberdeen
  - 1199.32.44003 Boehringer Ingelheim Investigational Site, Birmingham
  - 1199.32.44005 Boehringer Ingelheim Investigational Site, Birmingham
  - 1199.32.44009 Boehringer Ingelheim Investigational Site, Leeds
  - 1199.32.44004 Boehringer Ingelheim Investigational Site, Liverpool
  - 1199.32.44002 Boehringer Ingelheim Investigational Site, London
  - 1199.32.44008 Boehringer Ingelheim Investigational Site, Oxford
  - 1199.32.44001 Boehringer Ingelheim Investigational Site, Westbury on Trym

REFERENCES:
- [Derived] Glaspole I, Bonella F, Bargagli E, Glassberg MK, Caro F, Stansen W, Quaresma M, Orsatti L, Bendstrup E. Efficacy and safety of nintedanib in patients with idiopathic pulmonary fibrosis who are elderly or have comorbidities. Respir Res. 2021 Apr 26;22(1):125. doi: 10.1186/s12931-021-01695-y. PMID 33902584
- [Derived] Jouneau S, Crestani B, Thibault R, Lederlin M, Vernhet L, Valenzuela C, Wijsenbeek M, Kreuter M, Stansen W, Quaresma M, Cottin V. Analysis of body mass index, weight loss and progression of idiopathic pulmonary fibrosis. Respir Res. 2020 Nov 25;21(1):312. doi: 10.1186/s12931-020-01528-4. PMID 33239000
- [Derived] Brown KK, Martinez FJ, Walsh SLF, Thannickal VJ, Prasse A, Schlenker-Herceg R, Goeldner RG, Clerisme-Beaty E, Tetzlaff K, Cottin V, Wells AU. The natural history of progressive fibrosing interstitial lung diseases. Eur Respir J. 2020 Jun 25;55(6):2000085. doi: 10.1183/13993003.00085-2020. Print 2020 Jun. PMID 32217654
- [Derived] Richeldi L, Kolb M, Jouneau S, Wuyts WA, Schinzel B, Stowasser S, Quaresma M, Raghu G. Efficacy and safety of nintedanib in patients with advanced idiopathic pulmonary fibrosis. BMC Pulm Med. 2020 Jan 8;20(1):3. doi: 10.1186/s12890-019-1030-4. PMID 31914963
- [Derived] Kreuter M, Koegler H, Trampisch M, Geier S, Richeldi L. Differing severities of acute exacerbations of idiopathic pulmonary fibrosis (IPF): insights from the INPULSIS(R) trials. Respir Res. 2019 Apr 11;20(1):71. doi: 10.1186/s12931-019-1037-7. PMID 30971229
- [Derived] Xu Z, Li H, Wen F, Bai C, Chen P, Fan F, Hu N, Stowasser S, Kang J. Subgroup Analysis for Chinese Patients Included in the INPULSIS(R) Trials on Nintedanib in Idiopathic Pulmonary Fibrosis. Adv Ther. 2019 Mar;36(3):621-631. doi: 10.1007/s12325-019-0887-1. Epub 2019 Feb 7. PMID 30729456
- [Derived] Costabel U, Behr J, Crestani B, Stansen W, Schlenker-Herceg R, Stowasser S, Raghu G. Anti-acid therapy in idiopathic pulmonary fibrosis: insights from the INPULSIS(R) trials. Respir Res. 2018 Sep 3;19(1):167. doi: 10.1186/s12931-018-0866-0. PMID 30176872
- [Derived] Collard HR, Richeldi L, Kim DS, Taniguchi H, Tschoepe I, Luisetti M, Roman J, Tino G, Schlenker-Herceg R, Hallmann C, du Bois RM. Acute exacerbations in the INPULSIS trials of nintedanib in idiopathic pulmonary fibrosis. Eur Respir J. 2017 May 19;49(5):1601339. doi: 10.1183/13993003.01339-2016. Print 2017 May. PMID 28526798
- [Derived] Paterniti MO, Bi Y, Rekic D, Wang Y, Karimi-Shah BA, Chowdhury BA. Acute Exacerbation and Decline in Forced Vital Capacity Are Associated with Increased Mortality in Idiopathic Pulmonary Fibrosis. Ann Am Thorac Soc. 2017 Sep;14(9):1395-1402. doi: 10.1513/AnnalsATS.201606-458OC. PMID 28388260
- [Derived] Rinciog C, Watkins M, Chang S, Maher TM, LeReun C, Esser D, Diamantopoulos A. A Cost-Effectiveness Analysis of Nintedanib in Idiopathic Pulmonary Fibrosis in the UK. Pharmacoeconomics. 2017 Apr;35(4):479-491. doi: 10.1007/s40273-016-0480-2. PMID 28039616
- [Derived] Kolb M, Richeldi L, Behr J, Maher TM, Tang W, Stowasser S, Hallmann C, du Bois RM. Nintedanib in patients with idiopathic pulmonary fibrosis and preserved lung volume. Thorax. 2017 Apr;72(4):340-346. doi: 10.1136/thoraxjnl-2016-208710. Epub 2016 Sep 26. PMID 27672117
- [Derived] Corte T, Bonella F, Crestani B, Demedts MG, Richeldi L, Coeck C, Pelling K, Quaresma M, Lasky JA. Safety, tolerability and appropriate use of nintedanib in idiopathic pulmonary fibrosis. Respir Res. 2015 Sep 24;16:116. doi: 10.1186/s12931-015-0276-5. PMID 26400368
- [Derived] Richeldi L, du Bois RM, Raghu G, Azuma A, Brown KK, Costabel U, Cottin V, Flaherty KR, Hansell DM, Inoue Y, Kim DS, Kolb M, Nicholson AG, Noble PW, Selman M, Taniguchi H, Brun M, Le Maulf F, Girard M, Stowasser S, Schlenker-Herceg R, Disse B, Collard HR; INPULSIS Trial Investigators. Efficacy and safety of nintedanib in idiopathic pulmonary fibrosis. N Engl J Med. 2014 May 29;370(22):2071-82. doi: 10.1056/NEJMoa1402584. Epub 2014 May 18. PMID 24836310
- [Derived] Richeldi L, Cottin V, Flaherty KR, Kolb M, Inoue Y, Raghu G, Taniguchi H, Hansell DM, Nicholson AG, Le Maulf F, Stowasser S, Collard HR. Design of the INPULSIS trials: two phase 3 trials of nintedanib in patients with idiopathic pulmonary fibrosis. Respir Med. 2014 Jul;108(7):1023-30. doi: 10.1016/j.rmed.2014.04.011. Epub 2014 Apr 29. PMID 24834811

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Oral administration of placebo matching nintedanib soft gelatine capsules
- Nintedanib 150mg Bid: Oral administration of soft gelatine capsules of nintedanib 150mg twice daily (bid).
  Dose interruption and reduction to 100 mg bid dose were allowed to manage adverse events.
Period: Overall Study
Arm/Group | Placebo | Nintedanib 150mg Bid
Started | 206 | 309
Completed | 174 | 260
Not Completed | 32 | 49
Not completed — Adverse Event | 15 | 25
Not completed — Non compliant with protocol | 2 | 0
Not completed — Consent withdrawn, not due to AE | 12 | 23
Not completed — Not treated | 2 | 0
Not completed — Reason other than those stated above | 1 | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS consisted of randomised patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Nintedanib 150mg Bid | Total
Number analyzed (Participants) | 204 | 309 | 513
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (8.2) | 66.9 (8.4) | 66.9 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 58 | 99
  Male | 163 | 251 | 414

OUTCOME MEASURES:

1. Primary Outcome: Annual Rate of Decline in Forced Vital Capacity (FVC) Over 52 Weeks
Description: Forced vital capacity (FVC) is the total amount of air exhaled during the lung function test.
  For this endpoint reported means represent the adjusted rate
Time Frame: 52 weeks
Population: TS (Only patients with observed cases (OC) values were analysed)
Measure: Mean (Standard Error); unit: mL/year
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 204 | 309
mL/year | -239.91 (18.709) | -114.65 (15.327)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 150mg Bid; Random coefficient regression with fixed effects for treatment, gender, age, height and random effect of patient specific intercept and time. A hierarchical procedure was used in order to demonstrate the superiority of nintedanib over placebo for one primary and two key secondary endpoints. The consecutive steps of the hierarchy were only considered if the previous step was significant at the one-sided 2.5% level and the results were in favour of nintedanib; Test type: Superiority or Other; p < 0.0001, Random coefficient regression — The objective of this trial was to assess the superiority of nintedanib 150 mg bid compared to placebo on the annual rate of decline in FVC; The Roger-Kenward approximation was used to estimate denominators degrees of freedom; Mean Difference (Final Values) = 125.26, 95% CI 2-sided [77.68 to 172.84], Standard Error of Mean 24.209 — Within-patient errors are modelled by an Unstructured variance-covariance matrix. Inter-individual variability is modelled by a Variance-components variance-covariance matrix Nintedanib 150 mg bid versus Placebo

2. Secondary Outcome: Change From Baseline in Saint-George's Respiratory Questionnaire (SGRQ) Total Score at 52 Weeks
Description: This is a key secondary endpoint.
  SGRQ is a health-related quality of life questionnaire divided into 3 components : symptoms, activity and impact.
  The total score (summed weights) can range from 0 to 100 with a lower score denoting a better health status.
  Means provided are the adjusted means based on all analyzed patients in the model (not only patients with a baseline and measurement at week 52).
Time Frame: baseline and 52 weeks
Population: TS (Only patients with observed cases (OC) values were analysed)
Measure: Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 200 | 289
points on a scale | 4.39 (0.960) | 4.34 (0.799)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 150mg Bid; Mixed Model for Repeated Measures (MMRM), with fixed effects for treatment, visit, treatment-by-visit, baseline SGRQ Total score, baseline SGRQ Total score-by-visit and random effect for patient; Test type: Superiority or Other; p = 0.9657, Mixed Models Analysis; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-2.50 to 2.40], Standard Error of Mean 1.248 — Within-patient errors are modelled by compound symmetry covariance matrix Nintedanib 150 mg bid versus Placebo

3. Secondary Outcome: Time to First Acute Idiopathic Pulmonary Fibrosis (IPF) Exacerbation
Description: Due to rare events, the median of time to event is not calculable, thus the percentages of patients with (IPF) exacerbation are reported and represented as a key secondary endpoint. An acute exacerbation (reported as an AE by the investigator) was defined as follows:
  Otherwise unexplained clinical features including all of the following:
  * Unexplained worsening or development of dyspnoea within 30 days
  * New diffuse pulmonary infiltrates on chest X-ray, and/or new HRCT parenchymal abnormalities with no pneumothorax or pleural effusion (new ground-glass opacities) since the last visit
  * Exclusion of infection as per routine clinical practice and microbiological studies
  * Exclusion of alternative causes as per routine clinical practice including left heart failure, pulmonary embolism and identifiable cause of acute lung injury.
  Failure is the proportion of patients with at least one acute IPF exacerbation over 52 weeks, based on all investigator-reported AEs .
Time Frame: 52 weeks
Population: Treated Set (Only patients with observed cases (OC) values were analysed)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 204 | 309
percentage of participants
  Failure | 5.4 | 6.1
  Censored | 94.6 | 93.9
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 150mg Bid; Hazard Ratio is based on a Cox´s regression model with terms for treatment, gender, age and height; Test type: Superiority or Other; p = 0.6728, Log Rank; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.54 to 2.42] — Nintedanib 150 mg bid versus Placebo

4. Secondary Outcome: Absolute Change From Baseline in Forced Vital Capacity (FVC) Over 52 Weeks
Description: Means provided are the adjusted means and are based on all analysed patients in the model (not only patients with a change from baseline to week 52).
Time Frame: Baseline and 52 weeks
Population: TS (Only patients with observed cases (OC) values were analysed)
Measure: Mean (Standard Error); unit: mL
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 204 | 307
mL | -205.00 (16.544) | -95.07 (14.375)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 150mg Bid; Based on Mixed Model for Repeated Measures (MMRM), with fixed effects for treatment, visit, gender, age, height, treatment-by-visit, baseline FVC, baseline FVC-by-visit and random effect for patient; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 109.93, 95% CI 2-sided [71.27 to 148.59], Standard Error of Mean 19.708 — Within-patient errors are modelled by compound symmetry covariance matrix. Nintedanib 150 mg bid versus Placebo

5. Secondary Outcome: Relative Change From Baseline in Forced Vital Capacity (FVC) Over 52 Weeks
Description: Percentage change from baseline in FVC over 52 weeks. Means provided are the adjusted means and are based on all analysed patients in the model (not only patients with a change from baseline to week 52).
Time Frame: Baseline and 52 weeks
Population: TS (Only patients with observed cases (OC) values were analysed)
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 204 | 307
percent change | -7.38 (0.633) | -3.36 (0.550)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 150mg Bid; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 4.02, 95% CI 2-sided [2.54 to 5.50], Standard Error of Mean 0.753 — Within-patient errors are modelled by compound symmetry covariance matrix. Nintedanib 150 mg bid versus Placebo

6. Secondary Outcome: Absolute Change From Baseline in Forced Vital Capacity (FVC) (% Predicted) Over 52 Weeks
Description: as for outcome 4
Time Frame: Baseline and 52 weeks
Population: TS (Only patients with observed cases (OC) values were analysed)
Measure: Mean (Standard Error); unit: % predicted
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 204 | 307
% predicted | -5.98 (0.474) | -2.76 (0.408)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 150mg Bid; Based on Mixed Model for Repeated Measures (MMRM), with fixed effects for treatment, visit, gender, age, height, treatment-by-visit, baseline FVC [%predicted], baseline FVC [%predicted]-by-visit and random effect for patient; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.22, 95% CI 2-sided [2.11 to 4.33], Standard Error of Mean 0.564 — Within-patient errors are modelled by compound symmetry covariance matrix. Nintedanib 150 mg bid versus Placebo

7. Secondary Outcome: Relative Change From Baseline in Forced Vital Capacity (FVC) (% Predicted) Over 52 Weeks
Description: Percentage change from baseline in FVC (% predicted) at 52 weeks. Means provided are the adjusted means and are based on all analysed patients in the model (not only patients with a change from baseline to week 52).
Time Frame: Baseline and 52 weeks
Population: TS (Only patients with observed cases (OC) values were analysed)
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 204 | 307
percent change | -7.32 (0.634) | -3.32 (0.547)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 150mg Bid; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 4.00, 95% CI 2-sided [2.52 to 5.48], Standard Error of Mean 0.753 — Within-patient errors are modelled by compound symmetry covariance matrix. Nintedanib 150 mg bid versus Placebo

8. Secondary Outcome: Absolute Categorical Change of FVC (% Predicted) by Categories Over 52 Weeks - 5% Threshold
Description: Absolute categorical change of FVC (% predicted) by categories over 52 weeks - 5% threshold (decrease by >5%, increase by >5%, and change within ≤5%).
Time Frame: Baseline and 52 weeks
Population: TS (for patients with change from baseline in FVC (%predicted) at Week 52)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 165 | 250
percentage of participants
  Decrease > 5% | 52.7 | 34.8
  Change within ≤ 5% | 41.2 | 54.0
  Increase > 5% | 6.1 | 11.2

9. Secondary Outcome: Absolute Categorical Change of FVC (% Predicted) by Categories Over 52 Weeks - 10% Threshold
Description: Absolute categorical change of FVC (% predicted) by categories over 52 weeks - 10% threshold (decrease by 10%, increase by >10%, and change within ≤10%)
Time Frame: Baseline and 52 weeks
Population: TS (for patients with change from baseline in FVC (%predicted) at Week 52)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 165 | 250
percentage of participants
  Decrease > 10% | 29.7 | 12.8
  Change within ≤10% | 69.1 | 84.4
  Increase > 10% | 1.2 | 2.8

10. Secondary Outcome: FVC Responders Using 10% Threshold at 52 Weeks
Description: FVC responders using 10% threshold at 52 weeks, defined as patients with absolute decline in FVC% predicted no greater than 10% and with an FVC evaluation at 52 weeks.
Time Frame: 52 weeks
Population: Treated Set (Only patients with observed cases (OC) values were analysed)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 204 | 309
percentage of participants | 56.86 [50.00 to 63.47] | 70.55 [65.24 to 75.36]
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 150mg Bid; Logistic regression with terms treatment, age, gender, height and baseline FVC % predicted; Test type: Superiority or Other; p = 0.0007, Regression, Logistic; Odds Ratio (OR) = 1.914, 95% CI 2-sided [1.32 to 2.79] — Nintedanib 150 mg bid versus Placebo

11. Secondary Outcome: Proportion of FVC Responders Using 5% Threshold at 52 Weeks
Description: Proportion of FVC responders using 5% threshold at 52 weeks, defined as patients with absolute decline in FVC% predicted no greater than 5% and with an FVC evaluation at 52 weeks.
Time Frame: 52 weeks
Population: Treated Set (Only patients with observed cases (OC) values were analysed)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 204 | 309
percentage of participants | 38.24 [31.84 to 45.06] | 52.75 [47.18 to 58.25]
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 150mg Bid; Logistic regression with terms treatment, age, gender, height and baseline FVC % predicted; Test type: Superiority or Other; p = 0.0010, Regression, Logistic; Odds Ratio (OR) = 1.847, 95% CI 2-sided [1.28 to 2.66] — Nintedanib 150 mg bid versus Placebo

12. Secondary Outcome: Proportion of SGRQ Responders at 52 Weeks: Patient Reported Outcomes (PROs)
Description: Proportion of SGRQ responders at 52 weeks
  Responders defined as <= -4 points change in change from baseline in SGRQ total score at 52 weeks.
Time Frame: Baseline and 52 weeks
Population: Treated Set (Only patients with observed cases (OC) values were analysed)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 204 | 309
percentage of participants | 24.02 [18.67 to 30.33] | 20.39 [16.27 to 25.23]
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 150mg Bid; Logistic regression with terms treatment, baseline SGRQ total score; Test type: Superiority or Other; p = 0.4298, Regression, Logistic; Odds Ratio (OR) = 0.840, 95% CI 2-sided [0.55 to 1.29] — Nintedanib 150 mg bid versus Placebo

13. Secondary Outcome: Change From Baseline in SGRQ Symptom Score at 52 Weeks: Patient Reported Outcomes (PROs)
Description: SGRQ Symptom score is a sub-component of SGRQ total score and is concerned with the effect of respiratory symptoms, their frequency and severity. This score calculated as summed weights ranges from 0 to 100 with lower score denoting a better symptom-related quality of life.
  Means presented are the adjusted means and are based on all analyzed patients in the model (not only patients with a baseline and measurement at week 52).
Time Frame: Baseline and 52 weeks
Population: Treated Set (Only patients with observed cases (OC) values were analysed)
Measure: Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 202 | 300
points on a scale | 3.89 (1.351) | 1.56 (1.104)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 150mg Bid; Mixed Model for Repeated Measures (MMRM), with fixed effects for treatment, visit, treatment-by-visit, baseline SGRQ Symptoms component, baseline SGRQ Symptoms component-by-visit and random effect for patient; Test type: Superiority or Other; p = 0.1832, Mixed Models Analysis; Mean Difference (Final Values) = -2.32, 95% CI 2-sided [-5.74 to 1.10], Standard Error of Mean 1.744 — Within-patient errors are modelled by compound symmetry covariance matrix. Nintedanib 150 mg bid versus Placebo

14. Secondary Outcome: Change From Baseline in SGRQ Impact Score at 52 Weeks (Points): Patient Reported Outcomes (PROs)
Description: SGRQ Impact score is a sub-component of SGRQ total score and covers a range of aspects concerned with social functioning and psychological disturbances resulting from airway disease. This score calculated as summed weights ranges from 0 to 100 with lower score denoting a better impact-related quality of life.
  Means presented are the adjusted means and are based on all analyzed patients in the model (not only patients with a baseline and measurement at week 52).
Time Frame: Baseline and 52 weeks
Population: Treated Set (Only patients with observed cases (OC) values were analysed)
Measure: Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 202 | 291
points on a scale | 4.01 (1.113) | 4.87 (0.923)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 150mg Bid; Mixed Model for Repeated Measures (MMRM), with fixed effects for treatment, visit, treatment-by-visit, baseline SGRQ impact component, baseline SGRQ Impact component-by-visit and random effect for patient; Test type: Superiority or Other; p = 0.5510, Mixed Models Analysis; Mean Difference (Final Values) = 0.86, 95% CI 2-sided [-1.97 to 3.70], Standard Error of Mean 1.446 — Within-patient error are modelled by compound symmetry covariance matrix Nintedanib 150 mg bid versus Placebo

15. Secondary Outcome: Change From Baseline in SGRQ Activity Score at 52 Weeks (Points): Patient Reported Outcomes (PROs)
Description: SGRQ Activity score is a sub-component of SGRQ total score and concerned with activities that cause or are limited by breathlessness. This score calculated as summed weights ranges from 0 to 100 with lower score denoting a better activity-related quality of life.
  Means presented are the adjusted means and are based on all analyzed patients in the model (not only patients with a baseline and measurement at week 52).
Time Frame: baseline and 52 weeks
Population: Treated Set (Only patients with observed cases (OC) values were analysed)
Measure: Mean (Standard Error); unit: points on scale
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 200 | 295
points on scale | 5.81 (1.103) | 4.62 (0.906)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 150mg Bid; Mixed Model for Repeated Measures (MMRM), with fixed effects for treatment, visit, treatment-by-visit, baseline SGRQ Activities component, baseline SGRQ Activities component-by-visit and random effect for patient; Test type: Superiority or Other; p = 0.4049, Mixed Models Analysis; Mean Difference (Final Values) = -1.19, 95% CI 2-sided [-3.99 to 1.61], Standard Error of Mean 1.427 — Within-patient errors are modelled by compound symmetry covariance matrix Nintedanib 150 mg bid versus Placebo

16. Secondary Outcome: Change From Baseline in Idiopathic Pulmonary Fibrosis (IPF) Specific Version of SGRQ (SGRQ-I) Total Score at 52 Weeks (Points): Patient Reported Outcomes (PROs)
Description: SGRQ-I is the IPF specific version of SGRQ comprises of selected items from the SGRQ divided into three components, Symptoms, Activity and Impact. Each component is scored separately. The weights for all items with a positive responses are summed and the weights from missed items are deducted from the maximum possible weight for the total score.
  The total score is calculated by dividing the summed weights from positive items in the questionnaire by maximum possible weight for all items in the questionnaire. The total score can range from 0 to 100 with a lower score denoting a better health-related quality of life. Change from baseline is calculated as the difference between total score at week 52 and total score at baseline as measured by the scale.
Time Frame: Baseline and 52 weeks
Population: Treated Set (Only patients with observed cases (OC) values were analysed)
Measure: Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 200 | 290
points on a scale | 5.08 (0.992) | 4.30 (0.824)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 150mg Bid; Mixed Model for Repeated Measures (MMRM), with fixed effects for treatment, visit, treatment-by-visit, baseline SGRQ-I Total score, baseline SGRQ-I Total score-by-visit and random effect for patient; Test type: Superiority or Other; p = 0.5446, Mixed Models Analysis; Mean Difference (Final Values) = -0.78, 95% CI 2-sided [-3.31 to 1.75], Standard Error of Mean 1.289 — Within-patient errors are modelled by compound symmetry covariance matrix. Nintedanib 150mg versus placebo

17. Secondary Outcome: Change From Baseline in Shortness of Breath Questionnaire (SOBQ) at 52 Weeks: Patient Reported Outcomes (PROs)
Description: Shortness of Breath Questionnaire measures the shortness of breath. It comprises of 24 items. Each item is scored on a scale between 0-5 where 5 represents maximal breathlessness. The responses to all items are summed up to provide the overall score that can range from 0 (best outcome) to 120 (worst outcome).
  Means presented are the adjusted means and are based on all analyzed patients in the model (not only patients with a baseline and measurement at week 52).
Time Frame: baseline and 52 weeks
Population: Treated Set (Only patients with observed cases (OC) values were analysed)
Measure: Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 178 | 267
points on a scale | 7.61 (1.376) | 6.73 (1.113)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 150mg Bid; Mixed Model for Repeated Measures (MMRM), with fixed effects for treatment, visit, treatment-by-visit, baseline SOBQ score, baseline SOBQ score-by-visit and random effect for patient; Test type: Superiority or Other; p = 0.6203, Mixed Models Analysis; Mean Difference (Final Values) = -0.88, 95% CI 2-sided [-4.35 to 2.60], Standard Error of Mean 1.770 — Within-patient errors are modelled by compound symmetry covariance matrix. Nintedanib 150mg versus placebo

18. Secondary Outcome: Change From Baseline in Cough Symptoms Score of the Cough and Sputum Assessment Questionnaire (CASA-Q) Score at 52 Weeks: Patient Reported Outcomes (PROs)
Description: The cough domains of the Cough and Sputum Assessment Questionnaire (CASAQ(CD)) assess the frequency and severity of cough and sputum and their impact on everyday life. It contains 4 domains cough/sputum symptom and impact with each scale ranging from 0 to 100 with lower scores indicating higher symptoms/impact levels (worst outcome).
  Means presented are the adjusted means and are based on all analyzed patients in the model (not only patients with a baseline and measurement at week 52).
Time Frame: Baseline and 52 weeks
Population: Treated Set (Only patients with observed cases (OC) values were analysed)
Measure: Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 202 | 302
points on a scale | -0.52 (1.400) | -0.76 (1.136)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 150mg Bid; Mixed Model for Repeated Measures (MMRM), with fixed effects for treatment, visit, treatment-by-visit, baseline CASA-Q Cough symptoms score, baseline CASA-Q Cough symptoms score-by-visit and random effect for patient; Test type: Superiority or Other; p = 0.8942, Mixed Models Analysis; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-3.78 to 3.30], Standard Error of Mean 1.803 — Within- patient errors are modelled by compound symmetry covariance matrix. Nintedanib 150 mg versus Placebo

19. Secondary Outcome: Change From Baseline in Cough Impact Score of the Cough and Sputum Assessment Questionnaire (CASA-Q) Score at 52 Weeks : Patient Reported Outcomes (PROs)
Description: The cough domains of the Cough and Sputum Assessment Questionnaire (CASA-Q) assess the frequency and severity of cough and sputum and their impact on everyday life. It contains 4 domains cough/sputum symptom and impact with each scale ranging from 0 to 100 with lower scores indicating higher symptoms/impact levels (worst outcome).
  Means presented are the adjusted means and are based on all analyzed patients in the model (not only patients with a baseline and measurement at week 52).
Time Frame: Baseline and 52 weeks
Population: Treated Set (Only patients with observed cases (OC) values were analysed)
Measure: Mean (Standard Error); unit: points on a scale
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 202 | 302
points on a scale | -4.00 (1.240) | -2.36 (1.006)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 150mg Bid; Mixed Model for Repeated Measures (MMRM), with fixed effects for treatment, visit, treatment-by-visit, baseline CASA-Q Cough impact score, baseline CASA-Q Cough impact score-by-visit and random effect for patient; Test type: Superiority or Other; p = 0.3042, Mixed Models Analysis; Mean Difference (Final Values) = 1.64, 95% CI 2-sided [-1.49 to 4.77], Standard Error of Mean 1.596 — Within-patient errors are modelled by compound symmetry covariance matrix Nintedanib 150 mg versus Placebo

20. Secondary Outcome: Proportion of Patient's Global Impression of Change (PGI-C) Responders at 52 Weeks: Patient Reported Outcomes (PROs)
Description: Patient's Global Impression of Change (PGI-C) responders are defined as 'Very much better'/ 'Much better'/ 'A little better'/ 'No change'.
Time Frame: 52 weeks
Population: Treated Set (Only patients with observed cases (OC) values were analysed)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 204 | 309
percentage of participants | 54.90 [48.05 to 61.58] | 60.84 [55.30 to 66.12]
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 150mg Bid; Logistic regression with term treatment; Test type: Superiority or Other; p = 0.1818, Regression, Logistic; Odds Ratio (OR) = 1.276, 95% CI 2-sided [0.89 to 1.83] — Nintedanib 150mg versus placebo

21. Secondary Outcome: Change From Baseline in EuroQol 5-Dimensional Quality of Life Questionnaire (EQ-5D) Health State up to 52 Weeks : Patient Reported Outcomes (PROs)
Description: The EuroQol 5-dimensional Health State is based on a visual analog scale (EQ-VAS) representing the general patient's health state labelled from 100 (best imaginable health state) to 0 (worst imaginable health state). A higher score indicating a better health state. Change from baseline is calculated as the difference between health state at week 12, 24 and 52 respectively and health state at baseline as measured by the scale.
Time Frame: baseline, 12 weeks, 24 weeks and 52 weeks
Population: Treated Set (Only patients with observed cases (OC) values were analysed)
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 203 | 306
points on a scale
  12 weeks (N= 194, 287) | 0.04 (15.46) | -1.75 (16.42)
  24 weeks (N= 190, 279) | -0.84 (15.37) | -0.74 (17.92)
  52 weeks (N=160, 247) | -5.88 (19.17) | -2.46 (18.92)

22. Secondary Outcome: Risk of an Acute IPF Exacerbation Over 52 Weeks
Description: The incidence rate of exacerbations (calculated as the number of patients with at least 1 acute IPF exacerbation divided by the total number of years at risk in years*100)
Time Frame: 52 weeks
Population: Treated Set (Only patients with observed cases (OC) values were analysed)
Measure: Number; unit: Participants/Year *100
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 204 | 309
Participants/Year *100 | 5.6 | 6.6
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 150mg Bid; The log of the risk ratio was assumed to follow a normal distribution with mean 0 and variance equal to the sum of the reciprocals of the number of patients with at least one exacerbation in each treatment arm; Test type: Superiority or Other; p = 0.6793, Normal distribution; Risk ratio was calculated as the ratio of risk of exacerbation in both treatment groups; Risk Ratio (RR) = 1.17, 95% CI 2-sided [0.56 to 2.46] — Nintedanib 150mg bid versus placebo

23. Secondary Outcome: Time to Death Over 52 Weeks
Description: Due to rare events, the median of time to event is not calculable, thus the percentages of patients who did or did not experienced death before or at 372 days after randomisation or last contact date (whichever occurs first) are reported.
  Failure is the proportion of patients who died over 52 weeks (373 days time-period) .
Time Frame: 52 weeks
Population: Treated Set (Only patients with observed cases (OC) values were analysed)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 204 | 309
percentage of participants
  Failure | 6.4 | 4.2
  Censored | 93.6 | 95.8
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 150mg Bid; Hazard ratio is based on a Cox´s regression model with terms for treatment, gender, age and height; Test type: Superiority or Other; p = 0.2880, Log Rank; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.29 to 1.36] — Nintedanib 150mg bid versus placebo

24. Secondary Outcome: Time to Death Due to Respiratory Cause Over 52 Weeks (Adjudicated)
Description: Due to rare events, the median of time to event is not calculable, thus the percentages of participants who did or did not experienced death due to respiratory causes before or at 372 days after randomisation or last contact date (whichever occurs first) are reported.
  Failure is the the proportion of patients who died due to respiratory causes over 52 weeks (373 days time-period).
Time Frame: 52 weeks
Population: Treated Set (Only patients with observed cases (OC) values were analysed)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 204 | 309
percentage of participants
  Failure | 4.9 | 3.2
  Censored | 95.1 | 96.8
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 150mg Bid; Hazard ratio is based on Cox´s regression model with terms for treatment, gender, age and height; Test type: Superiority or Other; p = 0.3515, Log Rank; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.25 to 1.47] — Nintedanib 150mg versus placebo

25. Secondary Outcome: Time to On-treatment Death
Description: Due to rare events, the median of time to event is not calculable, thus the percentages of participants who did or did not die before or at last trial medication intake + 28 days were censored at last trial medication intake + 28 days and reported.
  Failure is the the proportion of patients who died on-treatment.
Time Frame: 52 weeks
Population: Treated Set (Only patients with observed cases (OC) values were analysed)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 204 | 309
percentage of participants
  Failure | 4.4 | 2.6
  Censored | 95.6 | 97.4
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 150mg Bid; Hazard ratio is based on a Cox´s regression model with terms for treatment, gender, age and height; Test type: Superiority or Other; p = 0.4869, Log Rank; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.26 to 1.82] — Nintedanib 150mg bid versus placebo

26. Secondary Outcome: Time to Death or Lung Transplant Over 52 Weeks
Description: Due to rare events, the median of time to event is not calculable, thus the percentages of participants who did or did not experience event (death or lung transplant) before or at 372 days after randomisation or last contact date (whichever occurs first) are reported.
  Failure is the proportion of patients who died or had lung transplant over 52 weeks (373 days time-period).
Time Frame: 52 weeks
Population: Treated Set (Only patients with observed cases (OC) values were analysed)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 204 | 309
percentage of participants
  Failure | 6.9 | 5.2
  Censored | 93.1 | 94.8
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 150mg Bid; Hazard ratio is based on Cox´s regression model with terms for treatment, gender, age and height; Test type: Superiority or Other; p = 0.4430, Log Rank; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.36 to 1.51] — Nintedanib 150mg versus placebo

27. Secondary Outcome: Time to Death or Lung Transplant or Qualifying for Lung Transplant Over 52 Weeks.
Description: Due to rare events, the median of time to event is not calculable, thus the percentages of participants who did or did not experienced death or lung transplant or qualifying for lung transplant over 52 weeks are reported. A patient was considered qualifying for lung transplant by the investigator if he or she fulfilled the following criteria:
  FVC <45% predicted or Carbon monoxide diffusion capacity (DL(CO)) <30% pred or Oxygen saturation on pulse oximetry (SpO2) <88% at rest, at sea level (to be adapted for other heights).
  These criteria were evaluated by investigators judgement. Failure is the proportion of patients who died or had lung transplant or qualified for lung transplant over 52 weeks (373 days time-period).
Time Frame: 52 weeks
Population: Treated Set (Only patients with observed cases (OC) values were analysed)
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 204 | 309
percentage of participants
  Failure | 18.1 | 14.9
  Censored | 81.9 | 85.1
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 150mg Bid; Hazard ratio is based on Cox´s regression model with terms for treatment, gender, age and height; Test type: Superiority or Other; p = 0.3558, Log Rank; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.52 to 1.25] — Nintedanib 150mg bid versus placebo

28. Secondary Outcome: Change From Baseline in SpO2 (Oxygen Saturation, Expressed in Percent) at Rest up Over 52 Weeks
Description: Means presented are the adjusted means. Adjusted mean is based on all analyzed patients in the model (not only patients with a change from baseline to week 52)
Time Frame: Baseline and 52 weeks
Population: Treated Set (Only patients with observed cases (OC) values were analysed)
Measure: Mean (Standard Error); unit: percent of oxygen saturation
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 199 | 299
percent of oxygen saturation | -0.53 (0.150) | -0.24 (0.129)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 150mg Bid; Mixed Model for Repeated Measures (MMRM), with fixed effects for treatment, visit, gender, age, height, treatment-by-visit, baseline SpO2, baseline SpO2-by-visit and random effect for patient; Test type: Superiority or Other; p = 0.1138, Mixed Models Analysis; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [-0.07 to 0.64], Standard Error of Mean 0.181 — Within-patient errors are modelled by compound symmetry covariance matrix. Nintedanib 150mg bid versus placebo

29. Secondary Outcome: Change From Baseline in Carbon Monoxide Diffusion Capacity (DLCO) at Rest Over 52 Weeks
Description: as for outcome 4
Time Frame: Baseline and 52 weeks
Population: Treated Set (Only patients with observed cases (OC) values were analysed)
Measure: Mean (Standard Error); unit: mmol/min/kPa
Arm/Group | Placebo | Nintedanib 150mg Bid
Number analyzed (Participants) | 195 | 286
mmol/min/kPa | -0.365 (0.0750) | -0.380 (0.0644)
Statistical Analysis 1: Comparison: Placebo vs Nintedanib 150mg Bid; Mixed Model for Repeated Measures with fixed effects for treatment, visit, gender, age, height, treatment-by-visit, baseline DLCO (HGB Corrected) [mmol/min/kPa], baseline DLCO (HGB Corrected) [mmol/min/kPa]-by-visit and random effect for patient; Test type: Superiority or Other; p = 0.8650, Mixed Models Analysis; Mean Difference (Final Values) = -0.015, 95% CI 2-sided [-0.191 to 0.161], Standard Error of Mean 0.0896 — Within-patient errors are modelled by compound symmetry covariance matrix. Nintedanib 150mg bid versus placebo

ADVERSE EVENTS:
Time Frame: From the first drug administration until 28 days after the last drug administration, up to 425 days
Groups:
- Nintedanib 150mg Bid: Oral administration of soft gelatine capsules of Nintedanib 150 mg twice daily (bid). Dose interruption and reduction to 100 mg bid dose were allowed to manage adverse events.
Arm/Group | Placebo | Nintedanib 150mg Bid
Serious Adverse Events (participants affected / at risk) | 55/204 | 96/309
Other Adverse Events (participants affected / at risk) | 177/204 | 289/309
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=204) | Nintedanib 150mg Bid (N=309)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 3
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiomegaly (Cardiac disorders) | 1 | 0
Cor pulmonale (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 3 | 1
Diastolic dysfunction (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 4
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Optic ischaemic neuropathy (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 2
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 2 | 5
General physical health deterioration (General disorders) | 0 | 1
Hyperthermia (General disorders) | 1 | 0
Impaired healing (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Polyp (General disorders) | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 2
Bronchitis (Infections and infestations) | 2 | 2
Bronchopneumonia (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
H1N1 influenza (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 3 | 1
Lung infection (Infections and infestations) | 0 | 2
Mycobacterial infection (Infections and infestations) | 0 | 1
Peritoneal abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 5 | 5
Pyelonephritis acute (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 2
Pulmonary function test decreased (Investigations) | 1 | 1
Weight decreased (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Balance disorder (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Motor dysfunction (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 3
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Glomerulonephritis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 3
Renal vasculitis (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 11 | 20
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1
Hypertensive crisis (Vascular disorders) | 1 | 2
Hypotension (Vascular disorders) | 0 | 1
Microscopic polyangiitis (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=204) | Nintedanib 150mg Bid (N=309)
Abdominal pain (Gastrointestinal disorders) | 2 | 26
Abdominal pain upper (Gastrointestinal disorders) | 9 | 23
Constipation (Gastrointestinal disorders) | 6 | 17
Diarrhoea (Gastrointestinal disorders) | 38 | 188
Flatulence (Gastrointestinal disorders) | 1 | 18
Nausea (Gastrointestinal disorders) | 12 | 70
Vomiting (Gastrointestinal disorders) | 4 | 39
Fatigue (General disorders) | 13 | 14
Bronchitis (Infections and infestations) | 27 | 35
Lower respiratory tract infection (Infections and infestations) | 11 | 16
Nasopharyngitis (Infections and infestations) | 34 | 39
Upper respiratory tract infection (Infections and infestations) | 18 | 28
Weight decreased (Investigations) | 12 | 24
Decreased appetite (Metabolism and nutrition disorders) | 14 | 26
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 17
Headache (Nervous system disorders) | 12 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 26 | 47
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 | 22
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 11 | 10
Rash (Skin and subcutaneous tissue disorders) | 6 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights